CLINICAL TRIAL: NCT06459726
Title: Effects of Shi Style Cervical Mobilization Versus Sustained Natural Apophyseal Glides on Pain,Strength and Functional Disability in Patients With Cervicogenic Headache.
Brief Title: Effects of Shi Style Cervical Mobilization Versus SNAGS in Patients With Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0182
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cervicogenic Headache
Keywords: muscle strength; manual therapy; unilateral headaches
MeSH Terms: conditions — Post-Traumatic Headache; Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shi style mobilisation (Active Comparator): In this group patient will receive Shi style cervical mobilization SCM including three crucial steps soothing tendon step, mobilization step and dredging collateral step 6 sessions over 2 weeks for 20 minutes.
  Interventions: Other: shi style mobilization
- SNAGS (Active Comparator): Patient will receive sustained natural apophyseal glides as described by brian mulligan. Patient position will be upright sitting when therapist will apply a sustained passive assesory glide while patient moves actively through available physiological range of motion in the direction in which symptoms are produced(25).
  the headache SNAG technique will be performed with the patient sitting on a chair in the erect posture. The therapist will handle C2 spinous process with the middle phalanx of one hand. With the other hand, he will perform ventral gliding on C2 for 10 repetitions holding for 10 seconds in each glide with a rest time of 30 seconds in between. Patient will be asked to report dizziness or any other symptom after procedure. If patient reports symptom then angle of application is changed to ensure symptom free treatment in all patients. Number of repetitions are increased gradually from 6 to 10 and end physiological movement is maintained for 10seconds
  Interventions: Other: SNAGS

INTERVENTIONS:
Other: shi style mobilization — Step 1 soothing tendon stepTherapist will aerate patient's neck 3 to 6 times.Step 2 moblization step Therapist will apply low velocity small amplitude oscillatory movement without thrust. Head will be in 45 degrees of flexion or extension. Repeat this for 3 to 6 times. Then distraction force is applied to the cervical. Step 3 dredging collateral step Therapist holds thenar and hypothenar muscles of patient's hand on affected side and gently shook the upper limb ebb and flow with small shaking and high frequency. Repeat the procedure 3 times 6 sesions over 2 weeks for 20minutes
  Arms: shi style mobilisation
Other: SNAGS — Patient will receive sustained natural apophyseal glides as described by brian mulligan. Patient position will be upright sitting when therapist will apply a sustained passive assesory glide while patient moves actively through available physiological range of motion in the direction in which symptoms are produced. the headache SNAG technique will be performed with the patient sitting on a chair in the erect posture. The therapist will handle C2 spinous process with the middle phalanx of one hand. With the other hand, he will perform ventral gliding on C2 for 10 repetitions holding for 10 seconds in each glide with a rest time of 30 seconds in between. Patient will be asked to report dizziness or any other symptom after procedure. If patient reports symptom then angle of application is changed to ensure symptom free treatment in all patientsNumber of repetitions are increased gradually from 6 to 10 and end physiological movement is maintained for 10second
  Arms: SNAGS

SUMMARY:
Cervicogenic headache (CGH) manifests as unilateral neck pain referred from the neck's soft tissues or bony structures. The aim of this study will be to compare the effectiveness of Shi style cervical mobilization versus Sustained Natural Apophyseal Glides on pain, strength and functional disability in patients with Cervicogenic Headache.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Jinnah hospital Lahore through consecutive sampling technique on 40 patients which will be allocated using simple random sampling through sealed opaque enveloped into Group A and Group B. Group A will be treated with shi style mobilizations with 6 sesions over 4 weeks for 20minutes. Group B will be treated with Sustained Natural Apophyseal Glides with Number of repetitions are increased gradually from 6 to 10 and end physiological movement is maintained for 10seconds. Outcome measures will be conducted through NPRS for pain , Deep Neck flexors strength by pressure Biofeedback, Dizziness Handicap Inventory for pain and change in dizziness, NDI for functional impairments and SF 36 for quality of life.Data will be analyzed through SPSS software version 25 .

ELIGIBILITY:
Inclusion Criteria:

* Age:18 to 65 years.
* Both male and females.
* Unilateral dominant headache.
* Positive International Headache Society Diagnostic Criteria (IHS) for cervicogenic headache.
* Decrease strength deep neck flexors by pressure biofeedback.
* Tenderness of the upper 3 cervical spine joints.

Exclusion Criteria:

* • Patients who received any treatment for CGH within the previous 3 months that would interfere with this study.

  * Pregnant females.
  * Inflammatory conditions in which manual therapy is contraindicated(29).
  * Cancer or brain diseases.
  * Recent fracture or injuries.
  * Congenital conditions of the cervical spine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
NPRS | 6th week
  Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain
Deep Neck flexors strength by pressure Biofeedback | 6th week
  Subjects will be positioned in supine lying, and the air unit of pressure biofeedback will be placed at the posterior aspect of the cervical spine just below the occiput and inflated to a baseline of 20 mmHg. They will be instructed to perform the cranio-cervical flexion movement such that the pressure rose to 22 mmHg and will hold this position for 10 seconds. A rest of 30 seconds will be provided, and the whole procedure will be repeated for 24, 26, 28, and 30 mmHg. Final reading will be taken when the subject is not able to hold the specific pressure for 10 seconds. Before the test, subjects will be given enough time to practice and examiner will observe for any substitution movements during the test. Test will be considered poor if subjects could not hold the position at 26 mmHg
Dizziness Handicap Inventory | 6th week
  The primary outcome will be the score on the Dizziness Handicap Inventory (DHI). The DHI Is a highly reliable and responsive tool. This questionnaire is validated and shows a high test-retest reliability (ICC = 0.98) he highest available score is 100, indicating the maximum level of self-perceived handicap (0-30 "low handicap", 30-60 "moderate handicap" and +60 "severe handicap")(32). The DHI consists of 25 items with 3 response levels that are categorized into subgroups as functional 36 points, emotional 36 points, and physical 28 points.
Quality of life SF36 | 6th week
  SF-36 was used to assess participants' health-related quality of life. It contains 36 questions divided into eight dimensions including physical functioning (10 items), role limitations due to physical health problems (four items), social functioning (two items), bodily pain (two items), general mental health (five items), vitality (four items), role limitations due to emotional health problems (three items), general health perceptions (five items), and reported health transition (one item). The score for each question will be the weight sum of the questions in each dimension. Physical (physical health, role physical, bodily pain, general health) and mental component summary scores (vitality, social functioning, role-emotional, and emotional well-being) were calculated(37). A total score can range from 0 to 100, where a higher score indicates better health status Assessments will be performed before, during, and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: rabbiya noor, phd, Principal Investigator — Study Principal Investigator
Locations (1):
- Jinnah Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yao M, Tang ZY, Cui XJ, Sun YL, Ye XL, Wang P, Zhong WH, Zhang RC, Li HY, Hu ZJ, Wang WM, Qiao WP, Li J, Gao Y, Shi Q, Wang YJ. Shi-Style Cervical Mobilizations Versus Massage for Cervical Vertigo: A Multicenter, Randomized, Controlled Clinical Trial. J Altern Complement Med. 2020 Jan;26(1):58-66. doi: 10.1089/acm.2019.0113. Epub 2019 Oct 3. PMID 31580705
- [Background] Nunez-Cabaleiro P, Leiros-Rodriguez R. Effectiveness of manual therapy in the treatment of cervicogenic headache: A systematic review. Headache. 2022 Mar;62(3):271-283. doi: 10.1111/head.14278. Epub 2022 Mar 16. PMID 35294051
- [Background] Cui XJ, Yao M, Ye XL, Wang P, Zhong WH, Zhang RC, Li HY, Hu ZJ, Tang ZY, Wang WM, Qiao WP, Sun YL, Li J, Gao Y, Shi Q, Wang Y. Shi-style cervical manipulations for cervical radiculopathy: A multicenter randomized-controlled clinical trial. Medicine (Baltimore). 2017 Aug;96(31):e7276. doi: 10.1097/MD.0000000000007276. PMID 28767566
- [Background] Haldeman S, Dagenais S. Cervicogenic headaches: a critical review. Spine J. 2001 Jan-Feb;1(1):31-46. doi: 10.1016/s1529-9430(01)00024-9. PMID 14588366
- [Background] Bogduk N. Cervicogenic headache: anatomic basis and pathophysiologic mechanisms. Curr Pain Headache Rep. 2001 Aug;5(4):382-6. doi: 10.1007/s11916-001-0029-7. PMID 11403743